CLINICAL TRIAL: NCT03650413
Title: A Phase II Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of UTTR1147A in Patients With Moderate to Severe Ulcerative Colitis or Crohn's Disease
Brief Title: An Extension Study to Evaluate the Long-Term Safety and Tolerability of UTTR1147A in Participants With Moderate to Severe Ulcerative Colitis or Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early by the Sponsor based on the interim analysis of Study GA39925 (NCT03558152) that showed low efficacy of UTTR1147A in ulcerative colitis. Development of the drug in this indication has been terminated.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA40209; 2017-004997-32 (EudraCT Number)
Record Dates: First submitted 2018-08-16; First posted 2018-08-28 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UTTR1147A (Experimental): All participants will have the opportunity to receive treatment with UTTR1147A until clinical remission is achieved. Participants will either receive treatment with UTTR1147A or undergo observation depending on disease status, as described in the protocol.
  Interventions: Drug: UTTR1147A

INTERVENTIONS:
Drug: UTTR1147A — UTTR1147A will be administered based on disease status, as described in the protocol.
  Other Names: Efmarodocokin alfa; RO7021610; RG7880; IL-22Fc

SUMMARY:
This study will evaluate the long-term safety and tolerability of UTTR1147A in participants with moderate to severe ulcerative colitis (UC) or Crohn's disease (CD), enrolling up to 320 participants from the parent studies: Phase Ib Study GA29469 (NCT02749630) and Phase II Study GA39925 (NCT03558152).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Study Entry:

* Prior enrollment in Study GA29469 or Study GA39925 and meeting protocol defined entry criteria

Inclusion Criteria for Study Entry and Study Re-Entry:

* Ability to comply with requirements of the study, in the investigator's judgment
* For women and men: use of highly effective contraception as defined by the protocol.

Exclusion Criteria:

Exclusion Criteria for Study Entry:

* Withdrawal of consent from parent study
* Discontinuation of study drug as required by the parent study protocol
* Discontinuation of study drug and withdrawal from Study GA29469 prior to Day 85 or from Study GA39925 prior to Week 8
* Noncompliance in the parent study, specifically defined as missing scheduled visits or non-adherence with background medications and concomitant medications

Exclusion Criteria for Study Entry and Study Re-Entry:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 8 weeks after the final dose of study drug or within 18 weeks after the final dose of study drug from GA39925, whichever is longer
* Any new malignancy, significant uncontrolled comorbidity, such as cardiac, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders, or signs or symptoms of infection judged by the investigator to be clinically significant since enrolling in the parent study
* Use of prohibited therapies as defined in the parent study
* Abnormal laboratory values, as defined in the protocol, recorded at the last visit in the parent study

Exclusion Criterion for Study Re-Entry:

* Use of prohibited concomitant therapy since enrolling in the extension study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (57):
- Carolina Digestive Diseases, Greenville, North Carolina, United States
- Bulgaria (2):
  - MHAT Saint Karidad EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment Hadji Dimitar OOD, Sliven
- LLC ARENSIA Exploratory Medicine, Tbilisi, Georgia
- Germany (4):
  - Gastroenterologische Spezialpraxis-Berlin-Karlshorst, Berlin
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitatsklinikum Schleswig Holstein; Klinik fur Allgemeine Innere Medizin, Kiel
  - St. Marien Krankenhaus; Med. Klinik, Ludwigshafen
- Greece (2):
  - Iatriko Palaiou Falirou; Gastrointestinal Department, Palaió Fáliro
  - EUROMEDICA General Clinic of Thessaloniki; Gastroenterology Department, Thessaloniki
- Portiuncula Hospital, Ballinasloe, Co Galway, Ireland
- Italy (4):
  - Complesso Integrato Columbus, Rome, Lazio
  - ASST di Monza - Azienda Ospedaliera San Gerardo; U.O. Farmacia -Settore A - Corpo Posteriore, Monza, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Azienda Ospedaliera Di Padova, Padua, Veneto
- ICS ARENSIA Exploratory Medicine, Chisinau, Moldova
- Poland (16):
  - SPZOZ Uniwersytecki SK nr 1 im N. Barlickiego UM w Lodzi; Oddz. Klin. Gastroenter. Og. i Onk., ?ód?
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy; Centrum Endoskopii Zabiegowej, Bydgoszcz
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Cz?stochowa
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gda?sk
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - ETG Kielce, Kielce
  - Gastromed SPK Niepubliczny Zaklad Opieki Zdrowotnej, Lublin
  - Klimed Marek Klimkiewicz, Piotrkow Trybunalski
  - Synexus - Poznan, Poznan
  - Clinical Research Center Sp. z o.o. MEDIC-R Spó?ka Komandytowa, Późna
  - Endoskopia Sp. z o.o., Sopot
  - Centrum Zdrowia MDM, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Przychodnia EuroMediCare, Wroc?aw
  - Melita Medical, Wroc?aw
  - Synexus - Wroclaw, Wroclaw
- Russia (4):
  - North-West State Medical University n.a. I.I. Mechnikov, Saint Petersburg, Sankt-Peterburg
  - Saint Martyr Elizabeth City Hospital, Saint Petersburg, Sankt-Peterburg
  - Irkutsk Research Centre Hospital of Siberian department of Russian Academy of Science, Irkutsk
  - Medical University Reaviz, Samara
- Serbia (6):
  - KBC Dr Dragisa Misovic Dedinje, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Clinical Center Kragujevac; Clinic Of Psychiatry, Kragujevac
  - General Hospital Vrsac, Vršac
  - Clinical Hospital Centre Zemun, Zemun
  - General Hospital Djordje Joanovic - Zrenjanin, Zrenjanin
- Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid, Spain
- Ukraine (13):
  - Regional Municipal Institution Chernivtsi Regional Clinical Hospital, Chernivtsi, Chernihiv Governorate
  - Medical Centre of PE First Private Clinic, Zhytomyr, Crimean Regional Governmenta
  - Ternopil University Hospital; Regional Center of Gastroenterology with Hepatology, Ternopil, Katerynoslav Governorate
  - Municipal Institution Zaporizhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporizhzhia, Kharkiv Governorate
  - Medical Center of LLC Medical Clinic Blagomed, Kyiv, KIEV Governorate
  - Medical Center of Limited Liability Company ?Harmoniya krasy?, Kyiv, KIEV Governorate
  - Medical Center of LLC Medical Center Dopomoga Plus, Kyiv, KIEV Governorate
  - Medical Center of Edelweiss Medics LLC, Kyiv, KIEV Governorate
  - Synexus Affiliate - MC of LLC Medbud-Clinic, Kyiv, KIEV Governorate
  - Med Center of International Institute of Clinical Trials LLC; Medical Center "OK!Clinic+", Kyiv, KIEV Governorate
  - Clinic of SRI of Invalid Rehab. (ESTC) of VNMU n.a. M.I.Pyrohov, Vinnytsia, Podolia Governorate
  - Transcarpathian Regional Clinical Hospital n.a. A. Novak; Rheumatology Department, Uzhhorod
  - Medical Center of Diaservice LLC; Division of clinical trials conduct, Department #3, Zaporizhzhia
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 143 patients were included in the intent-to-treat (ITT) population, with 128 patients allocated to study treatment and 15 patients that were not treated.
Pre-assignment Details: This is a single-arm open-label extension study. There is only one arm.
Groups:
- UTTR1147A: Participants enrolled in the extension study either received efmarodocokin alfa treatment (60 μg/kg intravenously [IV] every 4 weeks [Q4W]) or if they were in remission, underwent observation for up to 2 years (through Week 104), as determined based on the patient's disease status at the time of their last endoscopy in the parent study.
Period: Overall Study
Arm/Group | UTTR1147A
Started | 143
Completed | 82
Not Completed | 61
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 17
Not completed — Other | 9
Not completed — Physician Decision | 2
Not completed — Study Terminated By Sponsor | 16
Not completed — Withdrawal by Subject | 16

BASELINE CHARACTERISTICS:
Population: There was only 1 arm in this study. The protocol was written with this single group receiving treatment based upon remission status.
Arm/Group | UTTR1147A
Number analyzed (Participants) | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 135
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 142
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 142
  Not Stated | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 Scale (NCI CTCAE v4.0)
Time Frame: Up to 2 years
Population: The safety-evaluable population comprised 128 patients who received at least one dose of the study drug. There was only 1 arm in this open label extension study. Treatment was available to all study participants if they lost remission.
Measure: Count of Participants; unit: Participants
Arm/Group | UTTR1147A
Number analyzed (Participants) | 128
Participants
  Serious Adverse Events, Fatal SAEs and SAEs Related to Study Medication | 9
  Non-Serious Adverse Events Reported | 52

ADVERSE EVENTS:
Time Frame: From baseline up to 2 years
Description: The safety-evaluable population comprised 128 patients who received at least one dose of the study drug.There was only one arm of this study, however there was a subset of patients who received the IMP. This subset is defined here as the safety evaluable population.
Groups:
- UTTR1147A 60: Participants received treatment with UTTR1147A until clinical remission was achieved.
Arm/Group | UTTR1147A 60
All-Cause Mortality (participants affected / at risk) | 0/128
Serious Adverse Events (participants affected / at risk) | 9/128
Other Adverse Events (participants affected / at risk) | 52/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UTTR1147A 60 (N=128)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Amylase increased (Investigations) | 2 (2)
Lipase increased (Investigations) | 3 (4)
Venous thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UTTR1147A 60 (N=128)
Anaemia (Blood and lymphatic system disorders) | 15 (16)
COVID-19 (Infections and infestations) | 10 (11)
Headache (Nervous system disorders) | 8 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 30 (45)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT03650413/Prot_SAP_000.pdf